CLINICAL TRIAL: NCT02640807
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled Study of Two Dosing Frequencies of Recombinant Interleukin-7 (CYT107) Treatment to Restore Absolute Lymphocyte Counts in Sepsis Patients.
Brief Title: A Study of IL-7 to Restore Absolute Lymphocyte Counts in Sepsis Patients
Acronym: IRIS-7-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revimmune (Industry)
Collaborators: Vanderbilt University School of Medicine (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-107-15
Record Dates: First submitted 2015-12-14; First posted 2015-12-29 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2018-08

CONDITIONS: Severe Sepsis With Septic Shock
Keywords: sepsis lymphocytopenia IL-7; immune reconstitution
MeSH Terms: interventions — Interleukin-7; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- CYT107 high frequency (Experimental): Patients will receive Interleukin-7 (CYT107 liquid solution) at 10µg/kg twice a week for 4 weeks
  Interventions: Drug: Interleukin-7
- CYT107 low frequency (Experimental): Patients will receive Interleukin-7 (CYT107 liquid solution) at 10µg/kg twice a week for the first week, followed by CYT107 and Placebo once a week for the three following weeks
  Interventions: Drug: Interleukin-7; Drug: Placebo
- Control (Placebo Comparator): Patients will receive Placebo (NaCl 0.9%) twice a week for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interleukin-7 — IM (intra-muscular) administration of CYT107 recombinant glycosylated human IL-7 (SC administration for patients with INR (International Normalized Ratio) >2.5 or platelet count < 35,000
  Other Names: CYT107
  Arms: CYT107 high frequency; CYT107 low frequency
Drug: Placebo — IM administration of Placebo (SC administration for patients with INR>2.5 or platelet count < 35,000
  Other Names: NaCl 0.9%
  Arms: CYT107 low frequency; Control

SUMMARY:
A multicenter, randomized, double-blinded, placebo-controlled study of two dosing frequencies of recombinant Interleukin-7 (CYT107) treatment to restore absolute lymphocyte counts in sepsis patients; IRIS-7B (Immune Reconstitution of Immunosuppressed Sepsis patients).

A parallel study will be performed in France to allow a common statistical analysis of the primary end points and analysis for the enrolled patient population.

DETAILED DESCRIPTION:
Sepsis is the leading cause of death in critically ill patients in most intensive care units in Europe and the US. Recently, evidence has accumulated that sepsis progresses from a state of hyper-inflammation to a state of immunosuppression. This immunosuppressive phase is characterized by increased incidence of secondary infections often with relatively avirulent opportunistic type pathogens. Currently, new therapeutic approaches to sepsis are occurring using immuno-adjuvants that boost host immunity. One of the most promising agents Interleukin-7 is an essential, non-redundant, pluripotent cytokine produced mainly by bone marrow and thymic stromal cells that is required for T-cell survival.In addition to its anti-apoptotic properties, IL-7 induces potent proliferation of naïve and memory T-cells potentially supporting replenishment of the peripheral T-cell pool which is severely depleted during sepsis. These effects were confirmed in clinical trials at the National Cancer Institute and in HIV+ patients.

This clinical study will test the ability of IL-7 to restore the absolute lymphocyte counts in septic patients who have markedly reduced levels of circulating lymphocytes. An effect already confirmed in preclinical models of sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age ≥ 18 yrs and older but < 80 yrs
2. Patients with persistent suspected sepsis at 48-120 hrs after admission
3. Two or more criteria for the systemic inflammatory response syndrome (SIRS) (see reference #19 for SIRS criteria) and a clinically or microbiologically suspected infection.
4. At least one organ failure as defined by a SOFA (Sepsis-related organ failure assessment) score of ≥2 at any time point during the 48-120 hrs after admission to the ICU
5. Requirement of vasopressor treatment as follows: i) epinephrine or norepinephrine at ≥ 0.05 µg/kg/min ideal body weight; ii) vasopressin, or iii) dopamine at ≥ 4-5 μg/kg/min ideal body weight, continuously for 4 hrs or more, provided that at least 20 ml/kg of ideal body weight of crystalloid or an equivalent volume of colloid was administered during the 24-hour interval surrounding the start of vasopressor treatment, to maintain systolic pressure ≥ 90 mmHg or a mean arterial pressure ≥ 60 mmHg at any time point during their sepsis course preceding enrollment into the IL-7 study.
6. Lymphopenia with an absolute lymphocyte count ≤ 900 cells/mm3 at either the day of consent or the day prior to consent during their ICU stay.
7. Predicted length of stay in the ICU of up to two weeks after starting drug therapy treatment in the trial (ICU may also include a close medical ward on the same study site where the patient will remain under medical control of the Investigator).
8. Ability to obtain a signed informed consent from patient or LAR (Legally Authorized Representative) consent.

Exclusion Criteria:

1. Cancer with current chemotherapy or radiotherapy and/or .receipt of chemotherapy or radiotherapy within the last 6 weeks
2. Cardiopulmonary resuscitation within the previous 4 weeks without objective evidence of full neurologic recovery) or patients who have minimal chance of survival and are not expected to live > 3-5 days as defined by an APACHE II score of ≥ 35 at time of consideration for study eligibility
3. Patients with a history of or who currently have evidence of autoimmune disease including for example: myasthenia gravis, Guillain Barre syndrome, systemic lupus erythematosis, multiple sclerosis, scleroderma, ulcerative colitis, Crohn's disease, autoimmune hepatitis, Wegener's etc.
4. Patients who have received solid organ transplant or bone marrow transplant
5. Patients with active or a history of acute or chronic lymphocytic leukemia
6. AIDS-defining illness (category C) diagnosed within the last 12 months prior to study entry
7. History of splenectomy
8. Any hematologic disease associated with hypersplenism, such as thalassemia, hereditary spherocytosis, Gaucher's Disease, and autoimmune hemolytic anemia
9. Pregnant or lactating women
10. Participation in another investigational interventional study within the last 6 months prior to study entry, with the exception of studies aimed at testing sedation products belonging to standard of care such as Propofol, Dexmedetomidine, Midazolam.
11. Patients receiving immunosuppressive drugs, e.g., TNF-alpha inhibitors, for rheumatoid arthritis, inflammatory bowel disease or any other reason, or systemic corticosteroids other than hydrocortisone at a dose of 300 mg/day
12. Patients receiving concurrent immunotherapy or biologic agents including: growth factors, cytokines and interleukins, (other than the study medication); for example IL-2,growth factors, interferons, HIV vaccines, immunosuppressive drugs, hydroxyurea, immunoglobulins, adoptive cell therapy
13. Prisoners

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward SHERWOOD, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Richard HOTCHKISS, MD, PhD, Study Director — Washington University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hotchkiss RS, Moldawer LL. Parallels between cancer and infectious disease. N Engl J Med. 2014 Jul 24;371(4):380-3. doi: 10.1056/NEJMcibr1404664. No abstract available. PMID 25054723
- [Result] Hotchkiss RS, Karl IE. The pathophysiology and treatment of sepsis. N Engl J Med. 2003 Jan 9;348(2):138-50. doi: 10.1056/NEJMra021333. No abstract available. PMID 12519925
- [Result] Boomer JS, To K, Chang KC, Takasu O, Osborne DF, Walton AH, Bricker TL, Jarman SD 2nd, Kreisel D, Krupnick AS, Srivastava A, Swanson PE, Green JM, Hotchkiss RS. Immunosuppression in patients who die of sepsis and multiple organ failure. JAMA. 2011 Dec 21;306(23):2594-605. doi: 10.1001/jama.2011.1829. PMID 22187279
- [Result] Hall MW, Knatz NL, Vetterly C, Tomarello S, Wewers MD, Volk HD, Carcillo JA. Immunoparalysis and nosocomial infection in children with multiple organ dysfunction syndrome. Intensive Care Med. 2011 Mar;37(3):525-32. doi: 10.1007/s00134-010-2088-x. Epub 2010 Dec 10. PMID 21153402
- [Result] Hotchkiss RS, Coopersmith CM, McDunn JE, Ferguson TA. The sepsis seesaw: tilting toward immunosuppression. Nat Med. 2009 May;15(5):496-7. doi: 10.1038/nm0509-496. PMID 19424209
- [Result] Hotchkiss RS, Monneret G, Payen D. Immunosuppression in sepsis: a novel understanding of the disorder and a new therapeutic approach. Lancet Infect Dis. 2013 Mar;13(3):260-8. doi: 10.1016/S1473-3099(13)70001-X. PMID 23427891
- [Result] Hotchkiss RS, Monneret G, Payen D. Sepsis-induced immunosuppression: from cellular dysfunctions to immunotherapy. Nat Rev Immunol. 2013 Dec;13(12):862-74. doi: 10.1038/nri3552. Epub 2013 Nov 15. PMID 24232462
- [Result] Mackall CL, Fry TJ, Gress RE. Harnessing the biology of IL-7 for therapeutic application. Nat Rev Immunol. 2011 May;11(5):330-42. doi: 10.1038/nri2970. PMID 21508983
- [Result] Morre M, Beq S. Interleukin-7 and immune reconstitution in cancer patients: a new paradigm for dramatically increasing overall survival. Target Oncol. 2012 Mar;7(1):55-68. doi: 10.1007/s11523-012-0210-4. Epub 2012 Mar 2. PMID 22383042
- [Result] Unsinger J, Burnham CA, McDonough J, Morre M, Prakash PS, Caldwell CC, Dunne WM Jr, Hotchkiss RS. Interleukin-7 ameliorates immune dysfunction and improves survival in a 2-hit model of fungal sepsis. J Infect Dis. 2012 Aug 15;206(4):606-16. doi: 10.1093/infdis/jis383. Epub 2012 Jun 12. PMID 22693226
- [Result] Levy Y, Lacabaratz C, Weiss L, Viard JP, Goujard C, Lelievre JD, Boue F, Molina JM, Rouzioux C, Avettand-Fenoel V, Croughs T, Beq S, Thiebaut R, Chene G, Morre M, Delfraissy JF. Enhanced T cell recovery in HIV-1-infected adults through IL-7 treatment. J Clin Invest. 2009 Apr;119(4):997-1007. doi: 10.1172/JCI38052. Epub 2009 Mar 16. PMID 19287090
- [Derived] Francois B, Jeannet R, Daix T, Walton AH, Shotwell MS, Unsinger J, Monneret G, Rimmele T, Blood T, Morre M, Gregoire A, Mayo GA, Blood J, Durum SK, Sherwood ER, Hotchkiss RS. Interleukin-7 restores lymphocytes in septic shock: the IRIS-7 randomized clinical trial. JCI Insight. 2018 Mar 8;3(5):e98960. doi: 10.1172/jci.insight.98960. PMID 29515037

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CYT107 High Frequency | CYT107 Low Frequency | Control
Started | 9 | 8 | 10
Completed | 9 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYT107 High Frequency | CYT107 Low Frequency | Control | Total
Number analyzed (Participants) | 9 | 8 | 10 | 27
Age, Continuous [Mean (Full Range); unit: years] | 62 [33 to 80] | 68 [56 to 82] | 56 [33 to 77] | 62 [33 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 7 | 6 | 8 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 11
  France | 5 | 5 | 6 | 16
SOFA Score [Mean (Full Range); unit: units on a scale] — Sequential Organ Failure Assessment (SOFA) Score. Used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. The score can range from 0 - 24. High values indicate worse outcome.
  Ref:
  APA Vincent, et al. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units Critical Care Medicine: 1998; 26(11), 1793-1800.
  units on a scale | 6 [1 to 11] | 5 [1 to 9] | 8 [0 to 16] | 6 [0 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Immune Reconstitution of Lymphocytopenic Sepsis Patients
Description: Number of patients showing an increase of Absolute Lymphocyte Count >50% from baseline at Day 42.
  Kinetic of immune restoration through weekly measures of Absolute Lymphocyte Counts
Time Frame: Day 0 to 42
Measure: Count of Participants; unit: Participants
Arm/Group | CYT107 High Frequency | CYT107 Low Frequency | Control
Number analyzed (Participants) | 9 | 8 | 10
Participants | 8 | 7 | 8

2. Secondary Outcome: CYT107 Effect on Absolute Lymphocyte Count
Description: Number of Patients with Absolute Lymphocyte Count > 1.2 at Day 42
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | CYT107 High Frequency | CYT107 Low Frequency | Control
Number analyzed (Participants) | 7 | 6 | 7
Participants | 6 | 6 | 4

3. Secondary Outcome: CYT107 Immunogenicity
Description: number of patients with binding or neutralizing antibodies against CYT107 at Day 60
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | CYT107 High Frequency | CYT107 Low Frequency | Control
Number analyzed (Participants) | 9 | 8 | 10
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the treatment period (Days 1-28) and through to the end of the follow-up period (Day 42).
Arm/Group | CYT107 High Frequency | CYT107 Low Frequency | Control
All-Cause Mortality (participants affected / at risk) | 3/9 | 1/8 | 2/10
Serious Adverse Events (participants affected / at risk) | 7/9 | 4/8 | 5/10
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYT107 High Frequency (N=9) | CYT107 Low Frequency (N=8) | Control (N=10)
Lung Abscess (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute hypoxic event (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Papilledema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Relapse of endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ischemic Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophago-bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Bile leak (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Recurrent septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal collections (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Evisceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anastomotic leak (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Multi organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Septic embolism (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bowel perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toxic megacolon (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wound abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Empyema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYT107 High Frequency (N=9) | CYT107 Low Frequency (N=8) | Control (N=10)
Lung Abscess (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute hypoxic event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Persisting Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholestatis (Investigations) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 3 (3)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 4 (7) | 4 (6) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Weaning failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hemorrhagic gastric ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hypercapnic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ischemic colitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Cardiac disorders) | 2 (4) | 1 (1) | 1 (1)
High sodium (Investigations) | 2 (2) | 0 (0) | 1 (1)
Supra ventricular tachycardia (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Yeast infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
High potassium (Investigations) | 2 (2) | 0 (0) | 1 (1)
Cutaneous rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
High alkaline phosphatase (Investigations) | 3 (3) | 0 (0) | 2 (2)
Low phosphate (Investigations) | 2 (2) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Pressure ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Hepatic cytolysis (Renal and urinary disorders) | 3 (4) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoglycemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Necrotizing fingers (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ileopsoas hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Low Calcium (Investigations) | 1 (1) | 2 (2) | 0 (0)
DRESS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Wound abscess (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration pneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Investigations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract colonization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
High amylase (Investigations) | 0 (0) | 1 (1) | 0 (0)
High lipase (Investigations) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic alkalosis (Investigations) | 0 (0) | 1 (1) | 1 (1)
Low potassium (Investigations) | 0 (0) | 1 (1) | 1 (1)
Cerebral sequelae of hypoglycemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hemorrhagic shock (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Post operative bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
GI discomfort (cramping/bloating) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Low Absolute Lymphocyte Count (Investigations) | 0 (0) | 0 (0) | 1 (1)
Low sodium (Investigations) | 0 (0) | 0 (0) | 2 (2)
High phosphorus (Investigations) | 0 (0) | 0 (0) | 1 (1)
Ventilator associated pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Empyema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Investigations) | 0 (0) | 0 (0) | 1 (1)
High BUN (Investigations) | 0 (0) | 0 (0) | 2 (2)
Thrombocytosis (Investigations) | 0 (0) | 0 (0) | 1 (1)
High phosphate (Investigations) | 0 (0) | 0 (0) | 1 (1)
High magnesium (Investigations) | 0 (0) | 0 (0) | 2 (2)
Coagulopathy/low platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Ileal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Exp wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Low BUN (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT02640807/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT02640807/SAP_001.pdf